CLINICAL TRIAL: NCT05570981
Title: A Comprehensive Evaluation of the Impact of ATP on Laryngeal Symptoms, Hypersensitivity and Function - an Observational Controlled Study
Brief Title: A Comprehensive Evaluation of the Impact of ATP on Laryngeal Symptoms, Hypersensitivity and Function
Acronym: MISP COUGH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Emil Walsted, Principal Investigator, Bispebjerg Hospital
Other Study IDs: H-21076805
Record Dates: First submitted 2022-09-14; First posted 2022-10-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Chronic Refractory Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Refractory Cough (CRC): Individuals with a diagnosis of chronic refractory cough
  Interventions: Diagnostic Test: Laryngeal sensitivity testing
- Healthy controls: Healthy control subjects matched to the CRC group by age and gender
  Interventions: Diagnostic Test: Laryngeal sensitivity testing

INTERVENTIONS:
Diagnostic Test: Laryngeal sensitivity testing — Direct stimulation of the laryngeal adductor reflex, measurement of laryngeal EMG and our capability to assess functional laryngeal response to an inhalational challenge with laryngoscopic techniques.

SUMMARY:
OBJECTIVES

* To deliver a comprehensive model of laryngeal assessment, evaluating both the sensory and motor components of upper airway control and to relate this to symptom disturbance.
* Determine if laryngeal control is altered by coughing and the impact of repeated coughing on overall laryngeal control and relaxation to its baseline state.
* Evaluate if cell damage and tissue inflammation (including exposure to ATP) modulates laryngeal hypersensitivity and function, by using a comprehensive array of test modalities.

AIM To utilise state-of-the-art comprehensive assessment tools to evaluate laryngeal hypersensitivity and function in a cohort of individuals with chronic refractory cough and control subjects. The test modalities utilise direct stimulation of the laryngeal adductor reflex, measurement of laryngeal EMG and assessment of functional laryngeal response to an inhalational challenge with laryngoscopic techniques.

HYPOTHESIS Physiological markers of laryngeal hypersensitivity and dysfunction are highly prevalent in patients with chronic refractory cough and manifestations are driven by ATP stimulation.

OUTCOME MEASURES Measurements of laryngeal symptomatology will be measured over a run-in period and during challenge testing. Laryngeal relaxation will be studied using our novel tracking software capability, combining endoscopic imaging and physiological measurements of diaphragm activation.

ELIGIBILITY:
Inclusion criteria (controls)

* Age ≥ 18 years
* Healthy - with no history of any medical conditions
* No history of asthma / allergies
* Normal spirometric indices
* Non smoker

Inclusion criteria (patients)

* Age ≥ 18 years
* Chronic cough as per ATS definition (>8 weeks duration)
* High symptom burden (i.e. Cough VAS >= 40 mm at the screening visit)
* Chest radiograph or CT within 3 years of the screening visit with no abnormalities considered to contribute to chronic cough
* For patients with asthma: a confirmed diagnosis of asthma on the basis of asthma symptoms and reversible airflow obstruction (BDR 200mls + 12% change post bronchodilator and/or positive bronchoprovocation test).

Exclusion criteria

* Current smoker or a smoking history of >10 pack years
* Asthma that is not well-controlled, as per international asthma guidelines as specified by Global Initiative for Asthma (GINA)
* Recent exacerbation of cough or asthma within 4 weeks of inclusion
* Pregnancy or childbearing potential and no contraceptive treatment
* Respiratory tract infection within 4 weeks of inclusion
* Currently taking any of the following medications:

  * ACE inhibitors and within 3 months of inclusion
  * Antitussives (opioids, pregabalin, gabapentin, amitriptyline, nortriptyline or over-the-counter medications) within 2 weeks of inclusion
  * Medical treatments for GORD, eosinophilic bronchitis or other cough related conditions, initiated or changed (i.e. not in a stable regimen) for 4 weeks prior to inclusion.
* Medical history of COPD or chronic bronchitis
* Medical conditions/history or other circumstances which, in the judgement of the investigator, could increase the risk of adverse events or bias the study results

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) with chronic refractory cough and age-/gender matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal decrease in glottic anterior angle (degrees) during challenge testing | Baseline measurement is taken immediately before beginning the challenge test. Minimal value is taken from continuously measured glottic anterior angle, from immediately after baseline measurement and until immediately after challenge testing
  The maximal decrease in glottic anterior angle during challenge testing
Maximal increase in glottic anterior angle (degrees) after challenge testing | During challenge testing and from immediately after challenge testing until 5 minutes after challenge testing
  The difference between the minimal glottic anterior angle observed during challenge testing and the maximal glottic anterior angle observed from immediately after challenge testing and until 5 minutes after challenge testing
Maximal laryngeal relaxation time (seconds) | At baseline, during challenge testing and from immediately after challenge testing until 5 minutes after challenge testing
  Maximum time for glottic angle to normalise (i.e. achieve a value equal to or above the value prior to sensory stimulus)
Change in laryngeal relaxation time (seconds) during challenge testing | At baseline and immediately after challenge testing
  Change in time for glottic angle to normalise (i.e. achieve a value equal to or above the value prior to sensory stimulus)
Change in laryngeal relaxation time (seconds) in recovery | Immediately after challenge testing and at 5 minutes after challenge testing
  Change in time for glottic angle to normalise (i.e. achieve a value equal to or above the value prior to sensory stimulus)

SECONDARY OUTCOMES:
Cough VAS (0-100 mm) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Cough VAS dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Cough count and frequency | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Cough count dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.

OTHER OUTCOMES:
Breathing frequency (1/minute) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Breathing frequency dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Breathing frequency variability (entropy, unitless) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Breathing frequency variability dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Tidal volume (Litres) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Tidal volume dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Tidal volume variability (entropy, unitless) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Tidal volume variability dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Diaphragm activation (Root Mean Square of EMG mcV in a rolling 50ms window centered at the measureing point) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Diaphragm activation dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Oesophageal pressure (cmH2O) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Oesophageal pressure dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Gastric pressure (cmH2O) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Gastric pressure dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Trans-diaphragmatic pressure (cmH2O) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
  This is a descriptive delineation of the ATP/Transdiaphragmatic pressure dose/response relationship. The measure is taken at multiple times (see Time Frame) and visualised graphically.
Single cough episode duration (seconds) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing
Single cough episode intensity VAS (0-100 mm) | At baseline, during challenge testing at minutes 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30 and 4:00 (from immediately after an administered dose of ATP and until 15 seconds after an administered dose) and immediately after challenge testing

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No